CLINICAL TRIAL: NCT00133692
Title: INternational VErapamil SR Trandolapril STudy
Brief Title: INVEST: INternational VErapamil SR Trandolapril STudy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INVEST
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2010-08

CONDITIONS: Hypertension; Coronary Artery Disease
Keywords: Hypertension; Coronary Artery Disease; INVEST; Diabetes; Verapamil SR; Trandolapril; Atenolol; HCTZ
MeSH Terms: conditions — Hypertension; Coronary Artery Disease; Diabetes Mellitus | interventions — Hydrochlorothiazide

INTERVENTIONS:
Drug: Verapamil SR/Trandolapril/Hydrochlorothiazide (HCTZ)
Drug: Atenolol/HCTZ/Trandolapril

SUMMARY:
Because blood pressure affects the heart, blood vessels, kidneys, and the entire body, it is important to keep it as normal as possible. There are several different ways to control blood pressure and to prevent or limit the development of heart disease due to high blood pressure. The purpose of this study is to compare two treatments to see how well they work and the difference in their side effects. One treatment includes the use of a calcium antagonist drug (Isoptin sustained release [SR] or Verapamil SR). The other treatment excludes the calcium antagonist and may include a non-calcium antagonist drug called a beta blocker (Tenormin or Atenolol). Both treatments may also include medication called angiotensin converting enzyme (ACE) inhibitors and water pills. None of the drugs in this study are experimental, they are all approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
INVEST is an investigator initiated international, prospective, randomized study comparing two pharmacotherapy strategies to control hypertension in ambulatory patients with coronary artery disease (CAD). One strategy, the calcium antagonist care strategy, centers on a calcium antagonist (verapamil SR) followed by addition of an ACE inhibitor (trandolapril) and then diuretic (hydrochlorothiazide) as needed to achieve target blood pressures (BP). The other strategy, the non-calcium antagonist care strategy, uses a beta-blocker (atenolol) followed by addition of low-dose diuretic and then an ACE inhibitor (trandolapril) as needed to reach target BP. In either strategy additional drugs can be added provided the calcium antagonist is retained in the calcium antagonist care strategy and calcium antagonists are omitted in the non-calcium antagonist care strategy.

The study is organized into 15 international regions with about 1,500 study investigators randomizing approximately 22,000 patients who will be treated for at least two years. The primary response variable is the occurrence of adverse outcome, defined as any of the following events: all cause mortality, nonfatal MI or nonfatal stroke. A number of secondary response variables, including newly diagnosed diabetes will also be evaluated.

The primary objective of this trial is to examine the hypothesis that the risk for adverse outcomes (all cause mortality, nonfatal MI or nonfatal stroke) in hypertensive patients with CAD is at least equivalent during treatment of hypertension with a calcium antagonist strategy when compared with a non-calcium antagonist strategy.

Unique features of INVEST are, in addition to its size and international scope, its design to mimic standard clinical practice and its all electronic online data entry, drug distribution system, study management system, and electronic physician compensation. This system will permit the entire trial to be conducted via the Internet. This design is believed to be a forerunner of clinical trials research for the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 50 to no upper limit
* Hypertension documented according to the 6th report of the Joint National Committee on Detection and Evaluation of the treatment of high BP (JNC VI) and the need for drug therapy (previously documented hypertension in patients currently taking antihypertensive agents is acceptable)
* Documented CAD (e.g., classic angina pectoris (stable angina pectoris; Heberden angina pectoris), myocardial infarction three or more months ago, abnormal coronary angiography, or concordant abnormalities on two different types of stress tests)
* Willingness to sign informed consent

Exclusion Criteria:

* Unstable angina, angioplasty, coronary artery bypass graft surgery (CABG) or stroke within one month. Patients taking beta blockers after myocardial infarction are excluded if study enrollment is planned within 12 months of myocardial infarction. No time limitation if not taking beta-blocker.
* Use of a ß-blocker within past two weeks
* Patients without a pacemaker and any of the following:

  * Sinus bradycardia (< 50 beats/min.)
  * Sick sinus syndrome
  * Atrioventricular (AV)-block of more than 1st degree
* Documented contraindication to verapamil; documented contraindication to both atenolol and hydrochlorothiazide
* Atrial fibrillation/flutter with Wolff-Parkinson-White (WPW)-Syndrome
* Severe heart failure (New York Heart Association [NYHA] IV).
* Concomitant illnesses (e.g., severe renal failure [Serum creatinine ≥4.0 mg/dl], severe hepatic failure or known cirrhosis, etc.) which may affect outcome variables or where life expectancy is two years or less or which are likely to require frequent hospitalizations and/or treatment adjustments.
* Patients with psychiatric, cognitive, or social (e.g., alcoholism, etc.) conditions that would interfere with giving consent or cooperating or remaining available for follow-up for two years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22000
Dates: Start 1997-09; Study Completion 2003-02

PRIMARY OUTCOMES:
First occurrence of death or nonfatal myocardial infarction (MI) or nonfatal stroke

SECONDARY OUTCOMES:
Death
Nonfatal MI
Nonfatal stroke
Newly diagnosed diabetes
BP control
Cancer
Gastrointestinal (GI) bleeding
Alzheimer's Disease
Parkinson's Disease
Cardiovascular (CV) hospitalizations
Quality of life
Compliance

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Reynolds NA, Wagstaff AJ, Keam SJ. Trandolapril/verapamil sustained release: a review of its use in the treatment of essential hypertension. Drugs. 2005;65(13):1893-914. doi: 10.2165/00003495-200565130-00011. PMID 16114984
- [Background] Pepine CJ, Cooper-Dehoff RM. Cardiovascular therapies and risk for development of diabetes. J Am Coll Cardiol. 2004 Aug 4;44(3):509-12. doi: 10.1016/j.jacc.2004.03.071. PMID 15358012
- [Background] Keltai M, Johnson JA, Kowey PR, Ried LD, Tueth M. INVEST substudies: design and patient characteristics. Clin Cardiol. 2001 Nov;24(11 Suppl):V9-11. doi: 10.1002/clc.4960241704. PMID 11712776
- [Background] Erdine S, Handberg EM, Kolb B. Characteristics of patients with coronary artery disease and hypertension: a report from INVEST. Clin Cardiol. 2001 Nov;24(11 Suppl):V6-8. doi: 10.1002/clc.4960241703. PMID 11712775
- [Background] Questions and answers related to the INternational VErapamil SR/trandolapril STudy (INVEST). Clin Cardiol. 2001 Nov;24(11 Suppl):V30. No abstract available. PMID 11712774
- [Background] Conti CR, Cooper-DeHoff RM. How will INVEST and other hypertension trials change clinical practice? Clin Cardiol. 2001 Nov;24(11 Suppl):V24-9. doi: 10.1002/clc.4960241708. PMID 11712773
- [Background] Marks R, Bristol H, Conlon M, Pepine CJ. Enhancing clinical trials on the internet: lessons from INVEST. Clin Cardiol. 2001 Nov;24(11 Suppl):V17-23. doi: 10.1002/clc.4960241707. PMID 11712772
- [Background] Cooper-DeHoff R, Handberg E, Heissenberg C, Johnson K. Electronic prescribing via the internet for a coronary artery disease and hypertension megatrial. Clin Cardiol. 2001 Nov;24(11 Suppl):V14-6. doi: 10.1002/clc.4960241706. PMID 11712771
- [Background] Kolloch RE. INVEST: results of combined strategies to control blood pressure. Clin Cardiol. 2001 Nov;24(11 Suppl):V12-3. doi: 10.1002/clc.4960241705. PMID 11712770
- [Background] Pepine CJ, Handberg EM. The vascular biology of hypertension and atherosclerosis and intervention with calcium antagonists and angiotensin-converting enzyme inhibitors. Clin Cardiol. 2001 Nov;24(11 Suppl):V1-5. doi: 10.1002/clc.4960241702. PMID 11712769
- [Background] Pepine CJ, Handberg-Thurmond E, Marks RG, Conlon M, Cooper-DeHoff R, Volkers P, Zellig P. Rationale and design of the International Verapamil SR/Trandolapril Study (INVEST): an Internet-based randomized trial in coronary artery disease patients with hypertension. J Am Coll Cardiol. 1998 Nov;32(5):1228-37. doi: 10.1016/s0735-1097(98)00423-9. PMID 9809930
- [Result] Cooper-DeHoff RM, Gong Y, Handberg EM, Bavry AA, Denardo SJ, Bakris GL, Pepine CJ. Tight blood pressure control and cardiovascular outcomes among hypertensive patients with diabetes and coronary artery disease. JAMA. 2010 Jul 7;304(1):61-8. doi: 10.1001/jama.2010.884. PMID 20606150
- [Result] Denardo SJ, Messerli FH, Gaxiola E, Aranda JM Jr, Cooper-Dehoff RM, Handberg EM, Gong Y, Champion A, Zhou Q, Pepine CJ. Coronary revascularization strategy and outcomes according to blood pressure (from the International Verapamil SR-Trandolapril Study [INVEST]). Am J Cardiol. 2010 Aug 15;106(4):498-503. doi: 10.1016/j.amjcard.2010.03.056. PMID 20691307
- [Result] Denardo SJ, Gong Y, Nichols WW, Messerli FH, Bavry AA, Cooper-Dehoff RM, Handberg EM, Champion A, Pepine CJ. Blood pressure and outcomes in very old hypertensive coronary artery disease patients: an INVEST substudy. Am J Med. 2010 Aug;123(8):719-26. doi: 10.1016/j.amjmed.2010.02.014. PMID 20670726
- [Result] Beitelshees AL, Navare H, Wang D, Gong Y, Wessel J, Moss JI, Langaee TY, Cooper-DeHoff RM, Sadee W, Pepine CJ, Schork NJ, Johnson JA. CACNA1C gene polymorphisms, cardiovascular disease outcomes, and treatment response. Circ Cardiovasc Genet. 2009 Aug;2(4):362-70. doi: 10.1161/CIRCGENETICS.109.857839. Epub 2009 Jun 3. PMID 20031608
- [Result] Cooper-DeHoff RM, Handberg EM, Mancia G, Zhou Q, Champion A, Legler UF, Pepine CJ. INVEST revisited: review of findings from the International Verapamil SR-Trandolapril Study. Expert Rev Cardiovasc Ther. 2009 Nov;7(11):1329-40. doi: 10.1586/erc.09.102. PMID 19900016
- [Result] Gong Y, Handberg EM, Gerhard T, Cooper-Dehoff RM, Ried LD, Johnson JA, Pepine CJ; INVEST Investigators. Systolic blood pressure and subjective well-being in patients with coronary artery disease. Clin Cardiol. 2009 Nov;32(11):627-32. doi: 10.1002/clc.20501. PMID 19711440
- [Result] Bangalore S, Messerli FH, Franklin SS, Mancia G, Champion A, Pepine CJ. Pulse pressure and risk of cardiovascular outcomes in patients with hypertension and coronary artery disease: an INternational VErapamil SR-trandolapril STudy (INVEST) analysis. Eur Heart J. 2009 Jun;30(11):1395-401. doi: 10.1093/eurheartj/ehp109. Epub 2009 Apr 7. PMID 19351690
- [Result] Denardo SJ, Messerli FH, Gaxiola E, Aranda JM Jr, Cooper-Dehoff RM, Handberg EM, Gong Y, Champion A, Zhou Q, Pepine CJ. Characteristics and outcomes of revascularized patients with hypertension: an international verapamil SR-trandolapril substudy. Hypertension. 2009 Apr;53(4):624-30. doi: 10.1161/HYPERTENSIONAHA.108.111542. Epub 2009 Feb 23. PMID 19237684
- [Result] Johnson AD, Gong Y, Wang D, Langaee TY, Shin J, Cooper-Dehoff RM, Schork NJ, Binkley P, Pepine CJ, Johnson JA, Sadee W. Promoter polymorphisms in ACE (angiotensin I-converting enzyme) associated with clinical outcomes in hypertension. Clin Pharmacol Ther. 2009 Jan;85(1):36-44. doi: 10.1038/clpt.2008.194. Epub 2008 Oct 22. PMID 18946466
- [Result] Bavry AA, Anderson RD, Gong Y, Denardo SJ, Cooper-Dehoff RM, Handberg EM, Pepine CJ. Outcomes Among hypertensive patients with concomitant peripheral and coronary artery disease: findings from the INternational VErapamil-SR/Trandolapril STudy. Hypertension. 2010 Jan;55(1):48-53. doi: 10.1161/HYPERTENSIONAHA.109.142240. Epub 2009 Dec 7. PMID 19996066
- [Result] Pacanowski MA, Gong Y, Cooper-Dehoff RM, Schork NJ, Shriver MD, Langaee TY, Pepine CJ, Johnson JA; INVEST Investigators. beta-adrenergic receptor gene polymorphisms and beta-blocker treatment outcomes in hypertension. Clin Pharmacol Ther. 2008 Dec;84(6):715-21. doi: 10.1038/clpt.2008.139. Epub 2008 Jul 9. PMID 18615004
- [Result] Gerhard T, Gong Y, Beitelshees AL, Mao X, Lobmeyer MT, Cooper-DeHoff RM, Langaee TY, Schork NJ, Shriver MD, Pepine CJ, Johnson JA; INVEST Investigators. Alpha-adducin polymorphism associated with increased risk of adverse cardiovascular outcomes: results from GENEtic Substudy of the INternational VErapamil SR-trandolapril STudy (INVEST-GENES). Am Heart J. 2008 Aug;156(2):397-404. doi: 10.1016/j.ahj.2008.03.007. Epub 2008 Jun 20. PMID 18657677
- [Result] Bangalore S, Messerli FH, Cohen JD, Bacher PH, Sleight P, Mancia G, Kowey P, Zhou Q, Champion A, Pepine CJ; INVEST Investigators. Verapamil-sustained release-based treatment strategy is equivalent to atenolol-based treatment strategy at reducing cardiovascular events in patients with prior myocardial infarction: an INternational VErapamil SR-Trandolapril (INVEST) substudy. Am Heart J. 2008 Aug;156(2):241-7. doi: 10.1016/j.ahj.2008.02.023. PMID 18657652
- [Result] Kolloch R, Legler UF, Champion A, Cooper-Dehoff RM, Handberg E, Zhou Q, Pepine CJ. Impact of resting heart rate on outcomes in hypertensive patients with coronary artery disease: findings from the INternational VErapamil-SR/trandolapril STudy (INVEST). Eur Heart J. 2008 May;29(10):1327-34. doi: 10.1093/eurheartj/ehn123. Epub 2008 Mar 29. PMID 18375982
- [Result] Coca A, Messerli FH, Benetos A, Zhou Q, Champion A, Cooper-DeHoff RM, Pepine CJ. Predicting stroke risk in hypertensive patients with coronary artery disease: a report from the INVEST. Stroke. 2008 Feb;39(2):343-8. doi: 10.1161/STROKEAHA.107.495465. Epub 2007 Dec 27. PMID 18162623
- [Result] Beitelshees AL, Gong Y, Wang D, Schork NJ, Cooper-Dehoff RM, Langaee TY, Shriver MD, Sadee W, Knot HJ, Pepine CJ, Johnson JA; INVEST Investigators. KCNMB1 genotype influences response to verapamil SR and adverse outcomes in the INternational VErapamil SR/Trandolapril STudy (INVEST). Pharmacogenet Genomics. 2007 Sep;17(9):719-29. doi: 10.1097/FPC.0b013e32810f2e3c. PMID 17700361
- [Result] Cooper-DeHoff RM, Zhou Q, Gaxiola E, Cangiano JL, Garcia-Barreto D, Handberg E, Pepine CJ; INVEST Investigators. Influence of Hispanic ethnicity on blood pressure control and cardiovascular outcomes in women with CAD and hypertension: findings from INVEST. J Womens Health (Larchmt). 2007 Jun;16(5):632-40. doi: 10.1089/jwh.2006.0086. PMID 17627399
- [Result] Messerli F, Frishman WH, Elliott WJ, Bacher PH, Pepine CJ. Antihypertensive properties of a high-dose combination of trandolapril and verapamil-SR. Blood Press Suppl. 2007 Mar;1:6-9. PMID 17566313
- [Result] Brunner M, Cooper-DeHoff RM, Gong Y, Karnes JH, Langaee TY, Pepine CJ, Johnson JA; INVEST Investigators. Factors influencing blood pressure response to trandolapril add-on therapy in patients taking verapamil SR (from the International Verapamil SR/Trandolapril [INVEST] Study). Am J Cardiol. 2007 Jun 1;99(11):1549-54. doi: 10.1016/j.amjcard.2007.01.029. Epub 2007 Apr 16. PMID 17531579
- [Result] Langaee TY, Gong Y, Yarandi HN, Katz DA, Cooper-DeHoff RM, Pepine CJ, Johnson JA. Association of CYP3A5 polymorphisms with hypertension and antihypertensive response to verapamil. Clin Pharmacol Ther. 2007 Mar;81(3):386-91. doi: 10.1038/sj.clpt.6100090. PMID 17339868
- [Result] Bakris GL, Cooper-Dehoff RM, Zhou Q, Kupfer S, Champion A, Pepine CJ; INVEST Investigators. Dual therapy in hypertensive patients with coronary artery disease: the role of calcium channel blockers and beta-blockers. Am J Cardiovasc Drugs. 2007;7 Suppl 1:25-9. doi: 10.2165/00129784-200707001-00004. PMID 19845074
- [Result] Mancia G, Messerli F, Bakris G, Zhou Q, Champion A, Pepine CJ. Blood pressure control and improved cardiovascular outcomes in the International Verapamil SR-Trandolapril Study. Hypertension. 2007 Aug;50(2):299-305. doi: 10.1161/HYPERTENSIONAHA.107.090290. Epub 2007 Jul 2. PMID 17606861
- [Result] Uretsky S, Messerli FH, Bangalore S, Champion A, Cooper-Dehoff RM, Zhou Q, Pepine CJ. Obesity paradox in patients with hypertension and coronary artery disease. Am J Med. 2007 Oct;120(10):863-70. doi: 10.1016/j.amjmed.2007.05.011. PMID 17904457
- [Result] Cooper-Dehoff R, Cohen JD, Bakris GL, Messerli FH, Erdine S, Hewkin AC, Kupfer S, Pepine CJ; INVEST Investigators. Predictors of development of diabetes mellitus in patients with coronary artery disease taking antihypertensive medications (findings from the INternational VErapamil SR-Trandolapril STudy [INVEST]). Am J Cardiol. 2006 Oct 1;98(7):890-4. doi: 10.1016/j.amjcard.2006.04.030. Epub 2006 Aug 7. PMID 16996868
- [Result] Messerli FH, Mancia G, Conti CR, Hewkin AC, Kupfer S, Champion A, Kolloch R, Benetos A, Pepine CJ. Dogma disputed: can aggressively lowering blood pressure in hypertensive patients with coronary artery disease be dangerous? Ann Intern Med. 2006 Jun 20;144(12):884-93. doi: 10.7326/0003-4819-144-12-200606200-00005. PMID 16785477
- [Result] Cooper-DeHoff RM, Aranda JM Jr, Gaxiola E, Cangiano JL, Garcia-Barreto D, Conti CR, Hewkin A, Pepine CJ; INVEST Investigators. Blood pressure control and cardiovascular outcomes in high-risk Hispanic patients--findings from the International Verapamil SR/Trandolapril Study (INVEST). Am Heart J. 2006 May;151(5):1072-9. doi: 10.1016/j.ahj.2005.05.024. PMID 16644338
- [Result] Pepine CJ, Kowey PR, Kupfer S, Kolloch RE, Benetos A, Mancia G, Coca A, Cooper-DeHoff RM, Handberg E, Gaxiola E, Sleight P, Conti CR, Hewkin AC, Tavazzi L; INVEST Investigators. Predictors of adverse outcome among patients with hypertension and coronary artery disease. J Am Coll Cardiol. 2006 Feb 7;47(3):547-51. doi: 10.1016/j.jacc.2005.09.031. Epub 2006 Jan 18. PMID 16458134
- [Result] Ried LD, Tueth MJ, Taylor MD, Sauer BC, Lopez LM, Pepine CJ. Depressive symptoms in coronary artery disease patients after hypertension treatment. Ann Pharmacother. 2006 Apr;40(4):597-604. doi: 10.1345/aph.1G438. Epub 2006 Mar 28. PMID 16569807
- [Result] Elliott WJ, Hewkin AC, Kupfer S, Cooper-DeHoff R, Pepine CJ. A drug dose model for predicting clinical outcomes in hypertensive coronary disease patients. J Clin Hypertens (Greenwich). 2005 Nov;7(11):654-63. doi: 10.1111/j.1524-6175.2005.04800.x. PMID 16278523
- [Result] Zineh I, Cooper-Dehoff RM, Wessel TR, Arant CB, Sleight P, Geiser EA, Pepine CJ. Global differences in blood pressure control and clinical outcomes in the INternational VErapamil SR-Trandolapril STudy (INVEST). Clin Cardiol. 2005 Jul;28(7):321-8. doi: 10.1002/clc.4960280704. PMID 16075824
- [Result] Ried LD, Tueth MJ, Handberg E, Kupfer S, Pepine CJ; INVEST Study Group. A Study of Antihypertensive Drugs and Depressive Symptoms (SADD-Sx) in patients treated with a calcium antagonist versus an atenolol hypertension Treatment Strategy in the International Verapamil SR-Trandolapril Study (INVEST). Psychosom Med. 2005 May-Jun;67(3):398-406. doi: 10.1097/01.psy.0000160468.69451.7f. PMID 15911902
- [Result] Cooper-DeHoff RM, Handberg EM, Cohen J, Kowey P, Messerli FH, Mancia G, Cangiano JL, Gaxiola E, Garcia-Barreto D, Hewkin AC, Pepine CJ; INVEST Investigators. Characteristics of contemporary patients with hypertension and coronary artery disease. Clin Cardiol. 2004 Oct;27(10):571-6. doi: 10.1002/clc.4960271010. PMID 15553310
- [Result] Bakris GL, Gaxiola E, Messerli FH, Mancia G, Erdine S, Cooper-DeHoff R, Pepine CJ; INVEST Investigators. Clinical outcomes in the diabetes cohort of the INternational VErapamil SR-Trandolapril study. Hypertension. 2004 Nov;44(5):637-42. doi: 10.1161/01.HYP.0000143851.23721.26. Epub 2004 Sep 20. PMID 15381674
- [Result] Pepine CJ, Conti CR. Managing hypertension in European patients with coronary artery disease: design, results, and clinical implications of INVEST. Ital Heart J. 2004 Jun;5(6):411-6. No abstract available. PMID 15320564
- [Result] Brooks CS, Sowers JR. Importance of achieving lower blood pressure in hypertensive patients with diabetes. Hypertension. 2004 Nov;44(5):614-5. doi: 10.1161/01.HYP.0000143853.53256.f8. Epub 2004 Sep 13. No abstract available. PMID 15364899
- [Result] Pepine CJ, Handberg EM, Cooper-DeHoff RM, Marks RG, Kowey P, Messerli FH, Mancia G, Cangiano JL, Garcia-Barreto D, Keltai M, Erdine S, Bristol HA, Kolb HR, Bakris GL, Cohen JD, Parmley WW; INVEST Investigators. A calcium antagonist vs a non-calcium antagonist hypertension treatment strategy for patients with coronary artery disease. The International Verapamil-Trandolapril Study (INVEST): a randomized controlled trial. JAMA. 2003 Dec 3;290(21):2805-16. doi: 10.1001/jama.290.21.2805. PMID 14657064
- [Derived] Dasa O, Smith SM, Howard G, Cooper-DeHoff RM, Gong Y, Handberg E, Pepine CJ. Association of 1-Year Blood Pressure Variability With Long-term Mortality Among Adults With Coronary Artery Disease: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e218418. doi: 10.1001/jamanetworkopen.2021.8418. PMID 33914047
- [Derived] Elgendy IY, Bavry AA, Gong Y, Handberg EM, Cooper-DeHoff RM, Pepine CJ. Long-Term Mortality in Hypertensive Patients With Coronary Artery Disease: Results From the US Cohort of the International Verapamil (SR)/Trandolapril Study. Hypertension. 2016 Nov;68(5):1110-1114. doi: 10.1161/HYPERTENSIONAHA.116.07854. Epub 2016 Sep 12. PMID 27620390
- [Derived] Denardo SJ, Gong Y, Cooper-DeHoff RM, Farsang C, Keltai M, Szirmai L, Messerli FH, Bavry AA, Handberg EM, Mancia G, Pepine CJ. Effects of verapamil SR and atenolol on 24-hour blood pressure and heart rate in hypertension patients with coronary artery disease: an international verapamil SR-trandolapril ambulatory monitoring substudy. PLoS One. 2015 Apr 2;10(4):e0122726. doi: 10.1371/journal.pone.0122726. eCollection 2015. PMID 25835002
- [Derived] Bavry AA, Gong Y, Handberg EM, Cooper-DeHoff RM, Pepine CJ. Impact of aspirin according to type of stable coronary artery disease: insights from a large international cohort. Am J Med. 2015 Feb;128(2):137-43. doi: 10.1016/j.amjmed.2014.09.028. Epub 2014 Oct 15. PMID 25447610
- [Derived] Fontana V, McDonough CW, Gong Y, El Rouby NM, Sa AC, Taylor KD, Chen YD, Gums JG, Chapman AB, Turner ST, Pepine CJ, Johnson JA, Cooper-DeHoff RM. Large-scale gene-centric analysis identifies polymorphisms for resistant hypertension. J Am Heart Assoc. 2014 Nov 10;3(6):e001398. doi: 10.1161/JAHA.114.001398. PMID 25385345
- [Derived] Winchester DE, Cooper-Dehoff RM, Gong Y, Handberg EM, Pepine CJ; INVEST Investigators. Mortality implications of angina and blood pressure in hypertensive patients with coronary artery disease: New data from extended follow-up of the International Verapamil/Trandolapril Study (INVEST). Clin Cardiol. 2013 Aug;36(8):442-7. doi: 10.1002/clc.22145. Epub 2013 May 29. PMID 23720247
- [Derived] Gerhard T, Delaney JA, Cooper-Dehoff RM, Shuster J, Brumback BA, Johnson JA, Pepine CJ, Winterstein AG. Comparing marginal structural models to standard methods for estimating treatment effects of antihypertensive combination therapy. BMC Med Res Methodol. 2012 Aug 6;12:119. doi: 10.1186/1471-2288-12-119. PMID 22866767
- [Derived] Gong Y, Beitelshees AL, Cooper-DeHoff RM, Lobmeyer MT, Langaee TY, Wu J, Cresci S, Province MA, Spertus JA, Pepine CJ, Johnson JA. Chromosome 9p21 haplotypes and prognosis in white and black patients with coronary artery disease. Circ Cardiovasc Genet. 2011 Apr;4(2):169-78. doi: 10.1161/CIRCGENETICS.110.959296. Epub 2011 Mar 3. PMID 21372283
- [Derived] Niu Y, Gong Y, Langaee TY, Davis HM, Elewa H, Beitelshees AL, Moss JI, Cooper-Dehoff RM, Pepine CJ, Johnson JA. Genetic variation in the beta2 subunit of the voltage-gated calcium channel and pharmacogenetic association with adverse cardiovascular outcomes in the INternational VErapamil SR-Trandolapril STudy GENEtic Substudy (INVEST-GENES). Circ Cardiovasc Genet. 2010 Dec;3(6):548-55. doi: 10.1161/CIRCGENETICS.110.957654. PMID 21156931